CLINICAL TRIAL: NCT03616795
Title: Disposition of [14C]-LY3154207 Following Oral Administration in Healthy Male Subjects
Brief Title: Study of LY3154207 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16303; I7S-MC-HBEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — LY3154207

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3154207 and [14C]-LY3154207 (Experimental): A single dose of LY3154207 and [14C]-LY3154207administered orally.
  Interventions: Drug: LY3154207; Drug: [14C]-LY3154207

INTERVENTIONS:
Drug: LY3154207 — Administered orally
Drug: [14C]-LY3154207 — Administered orally

SUMMARY:
The main purpose of this study is to measure how much of the study drug gets into the bloodstream and how long it takes the body to get rid of it. This study will involve a single dose of 14C radiolabelled LY3154207. This means that a radioactive substance C14 will be incorporated into the study drug, to investigate the study drug and its breakdown products, to find out how much of these pass from blood into urine, feces and expired air. The study will last about 4 weeks. Screening is required within 28 days prior to the start of the study and follow up is required approximately 7 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 19 to 32.0 kilogram per meter square (kg/m²)
* Are 18 to 50 years old, inclusive, at the time of screening

Exclusion Criteria:

* Are currently or have been smokers or users of tobacco or nicotine replacement products within the 3 months prior to admission and/or have positive cotinine at screening or check-in
* Are unwilling to refrain from consuming caffeine- or xanthine-containing food and drink from 48 hours prior to admission and while resident in the CRU
* Have consumed grapefruits or grapefruit-containing products, Seville oranges or Seville orange-containing products, star fruits or star fruit-containing products within 7 days prior to dosing or intend to consume during the study
* Have participated in a [14C]-study within the last 4 to 6 months prior to admission for this study. The total 12-month exposure from this study and a maximum of 1 other previous [14C]-study within 6 to 12 months of this study (if the previous studies' radiation exposure is not known) or a maximum of 2 other previous [14C]-studies within 4 to 12 months of this study
* Have a history of clinically significant adverse drug reactions or "drug allergy" to more than 3 types of systemically administered medications (all penicillins and cephalosporins may be considered 1 type of medication for this purpose)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3154207 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered | Baseline through 552 hours after administration of study drug
  Urinary Excretion of LY3154207 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3154207 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered | Baseline through 552 hours after administration of study drug
  Fecal Excretion of LY3154207 Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY3154207 | Predose through 144 hours after administration of study drug
  Pharmacokinetics: Cmax of LY3154207
Pharmacokinetics: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC[0-∞]) | Predose through 144 hours after administration of study drug
  Pharmacokinetics: AUC(0-∞)
Total Number of Metabolites | Baseline through 552 hours after administration of study drug
  Total Number of Metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Wilbraham D, Biglan KM, Svensson KA, Tsai M, Kielbasa W. Safety, Tolerability, and Pharmacokinetics of Mevidalen (LY3154207), a Centrally Acting Dopamine D1 Receptor-Positive Allosteric Modulator (D1PAM), in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Apr;10(4):393-403. doi: 10.1002/cpdd.874. Epub 2020 Oct 7. PMID 33029934